CLINICAL TRIAL: NCT06677749
Title: Skeletal Muscle Myokine Response to Acute Eccentric Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 60484
Record Dates: First submitted 2024-07-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-07

CONDITIONS: Skeletal Muscle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eccentric Exercise (Experimental): 300 repetitions of isokinetic dynamometer eccentric knee extensions.
  Interventions: Procedure: Eccentric resistance-exercise

INTERVENTIONS:
Procedure: Eccentric resistance-exercise — Each participant will complete 300 repetitions of eccentric knee extensions using an isokinetic dynamometer after a baseline skeletal muscle biopsy is taken. Three hours following this, a second muscle biopsy will be taken to evaluate the changes in the dependent variables being measured (myokines).

SUMMARY:
The purpose of this study is to evaluate the acute local skeletal muscle inflammatory response to thigh muscle (quadriceps) eccentric muscle actions. Eccentric muscle actions occur when the muscle is lengthening as it contracts. This is a pilot project to assess the degree of inflammatory biomarkers, called myokines, that are released locally in skeletal muscle tissue after an acute bout of resistance-exercise using a resistance-exercise machine called an isokinetic dynamometer.

DETAILED DESCRIPTION:
The intervention will involve one session of maximal eccentric exercise of the knee extensor muscles (quadriceps) of the right leg. During the 24-hour period preceding the intervention, participants will be asked to refrain from any for of moderate-vigorous physical activity or exercise. Participants will perform 30 sets of 10 repetitions of maximal isokinetic eccentric knee extensions at 60 degrees/second with 1-minute of rest between each set. Before completing the exercise bout, each participant will be asked to remain in a seated position (resting) for 30-minutes and then provide a skeletal muscle biopsy using the modified Bergstrom with suction muscle biopsy technique from the vastus lateralis on the right leg. This will be done for the baseline assessment of 5 myokines including apelin, fibroblast growth factor-21, irisin, interleukin-6, and interleukin-15. Then the participants will complete the exercise bout as described above. They will then rest quietly in the laboratory for 3-hours and wait for the second skeletal muscle biopsy to be taken following this 3-hour wait.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* healthy
* recreationally active (>/= 150 minutes of moderate to vigorous physical activity per week for at least the past three months)

Exclusion Criteria:

* "yes" answer to the Get Active Questionnaire which screens for health conditions that may affect exercise ability

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Apelin | Baseline and 3-hours post-exercise
  Concentration of apelin in skeletal muscle tissue
Fibroblast growth factor-21 | Baseline and 3-hours post-exercise
  Concentration of fibroblast growth factor-21 in skeletal muscle tissue
Irisin | Baseline and 3-hours post-exercise
  Concentration of irisin in skeletal muscle tissue
Interleukin-6 | Baseline and 3-hours post-exercise
  Concentration of interleukin-6 in skeletal muscle tissue
Interleukin-15 | Baseline and 3-hours post-exercise
  Concentration of interleukin-15 in skeletal muscle tissue

SECONDARY OUTCOMES:
Body mass | Baseline
  Body mass in kilograms
Body height | Baseline
  Body height in meters
Body mass index | Baseline
  Body mass index in kg/m^2
Fat mass | Baseline
  Fat mass in kilograms
Fat free mass | Baseline
  Fat free mass in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Cornish, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Applied Research Centre, Faculty of Kinesiology, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No